CLINICAL TRIAL: NCT03810339
Title: A Phase II Open Label Study of Toripalimab, a PD-1 Antibody, in Participants With POLE or POLD-1 Mutated and Non-MSI-H Advanced Solid Tumors
Brief Title: Toripalimab as Monotherapy in Participants With POLE or POLD-1 Mutated and Non-MSI-H Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, President and Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPM
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor; Advanced Cancer
Keywords: Immune checkpoint inhibitor; POLE/POLD mutation; non-MSI-H
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab (Experimental): Toripalimab, 240mg, every 3 weeks until disease progress or intolerable toxicity
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab, 240mg, every 3 weeks until disease progress or intolerable toxicity

SUMMARY:
The purpose of this study is to evaluate the response of toripalimab (JS001), a PD1 antibody, in participants with POLE or POLD-mutated and non microsatellite instability (non-MSI-H) advanced solid cancers.

DETAILED DESCRIPTION:
Immune checkpoint inhibitor (ICI) therapy including antibodies targeting PD-1/PD-L1 or CTLA-4 has greatly advanced the cancer treatments. Recent studies have identified several predictive markers for ICI which includes microsatellite instability (MSI), PD-L1 expression and tumor mutation burden (TMB). DNA polymerase epsilon (POLE) and delta (POLD) are in charge of DNA replication as well as proofreading during DNA replication. Their germline or somatic mutations can lead to DNA repair deficiencies and carcinogenesis. The investigators has found that the POLE or POLD mutation causes an increased TMB in cancer patients and may lead to a better survival to ICI. Therefore, the purpose of this study is to evaluate the efficacy of toripalimab , a PD1 antibody, in participants with POLE or POLD-mutated and non microsatellite instability high (non-MSI-H) advanced solid cancers. This is a Phase II, open label, single arm study. Participants enrolled in this study received toripalimab 240mg, every 3 weeks until disease progress or intolerable toxicity. Primary endpoints is ORR and secondary endpoints are OS, PFS and safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants must provide written informed consent to participate
* Adult aged between 18 and 75 years old
* Participants with Histologically- or cytologically- proven advanced solid tumors and not responding to standard therapy
* MSS (microsatellite sability) or MSI-L (microsatellite instability-low) or pMMR status
* Germline mutations or somatic mutations in POLE or POLD (synonymous mutation is excluded)
* Patients refuse any conventional chemotherapy or targeted therapy
* Patients are willing to take biopsy of tumor tissue and take blood samples before treatment (blood samples are also taken at each time of therapeutic evaluation)
* Participants must have at least one measurable site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Lesions previously treated with radiotherapy should not be regarded as target lesions unless there is a definite progression of the lesion after radiotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Estimated life expectancy is greater than 3 months
* Participants can provide more than 10 paraffin sections of tumor tissue
* No history of radiotherapy or received non-targeted radiotherapy outside the target lesions for this study more than 4 weeks ago before the first dose of study treatment
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x (5 x in participants with liver metastasis) upper limit of normal (ULN)
* Albumin ≥ 3 g/dL
* Alkaline phosphatase ≤ 2.5 x ULN.
* Serum bilirubin <1.5 mg/dL
* Creatinine ≤ ULN.
* Absolute neutrophil count ≥ 1.5X10E9/L
* Platelets ≥ 100 x 10E9/L
* Hemoglobin ≥ 90 g/L
* For females of childbearing potential (defined as <2 years after last menstruation or not surgically sterile), a negative serum pregnancy test must be performed within 21 days of the first dose of study treatment.
* For females: agreement to contraception during the study treatment period and for at least 28 days after the last dose of study treatment

Exclusion Criteria:

* Patients with confirmed or suspected brain metastases
* Patients with cancerous meningitis
* Patients without germline mutations or somatic mutations in POLE and POLD
* MSI-H (microsatellite instability-high) or dMMR
* Prior treatment with PD-1 inhibitors, PD-L1 inhibitors or CTLA-4 inhibitors (or other inhibitors in T cell co-stimulatory signals or checkpoint pathways)
* Known history or evidence of cytotoxic drug therapy, biologic drug therapy (such as monoclonal antibodies), immunotherapy (such as interleukin 2 or interferon), or other investigational drugs therapy in the 4 weeks before the first dose of study treatment
* Known history or evidence of significant immunodeficiency (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, hyperthyroidism and hypothyroidism; Patients with vitiligo or asthma completely relieved can be included. Asthma that requires medical intervention cannot be included)
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisolone equivalent) or other immunosuppressive medications
* Patients with active tuberculosis. Known history of antituberculosis drugs treatment in 1 year before the first dose of study treatment
* Administration of an anti-infection vaccine (e.g. influenza vaccine, chickenpox vaccine) in the 4 weeks before the first dose of study treatment
* Symptomatic heart failure, coronary heart disease (CHD), myocardial infarction in the 6 months before the first dose of study treatment
* Known allergy to JS001 or its excipients
* Pregnant or breastfeeding females
* Other prior malignancy active within the previous 5 years except for non-melanoma skin cancer
* Persons without legal capacity
* Positive test for HIV or AIDS
* Positive test for HbsAg and HBV-DNA copy numbers (≥ 1000cps/ml)
* Positive test for HCV
* Any medical disorder or condition that, in the opinion of the investigator, may affect the compliance or the signing of informed consent, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rates (ORR) | up to 2 years
  the ratio of patients whose efficiency evaluation is CR or PR

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 2 years
  defined as the period from the first dose of study treatment to loss of follow-up or death
Progression free survival (PFS) | up to 2 years
  defined as the time from the first dose of study treatment to disease progression
Adverse Events (AEs) | up to 2 years
  All treatment-related adverse events (AEs) were categorized according to the National Cancer Institute's Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided